CLINICAL TRIAL: NCT00002235
Title: A Phase II, 48-Week, Open-Label Study Designed to Evaluate the Safety, Tolerability, and Efficacy of a Simplified Dosing Regimen of Viracept (Nelfinavir Mesylate) 1250 Mg BID, Crixivan (Indinavir Sulfate) 1200mg q12h, and Sustiva (Efavirenz; DMP-266) 600 Mg q24h for the Treatment of HIV-1 Infection in Non-Nucleoside Reverse Transcriptase Inhibitor and Protease Inhibitor Naive Patients
Brief Title: A Study on the Safety and Effectiveness of Twice-Daily Nelfinavir Plus Twice-Daily Indinavir Plus Efavirenz in HIV-Positive Patients Who Have Never Taken Non-Nucleoside Reverse Transcriptase Inhibitors (NNRTIs) or Protease Inhibitors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Collaborators: Agouron Pharmaceuticals (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Masking: None | Purpose: Treatment
Other Study IDs: 259G; ICC 602
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2000-03

CONDITIONS: HIV Infections
Keywords: Drug Therapy, Combination; HIV Protease Inhibitors; Indinavir; Nelfinavir; Reverse Transcriptase Inhibitors; Anti-HIV Agents; efavirenz
MeSH Terms: conditions — HIV Infections | interventions — Indinavir; Nelfinavir; efavirenz

INTERVENTIONS:
Drug: Indinavir sulfate
Drug: Nelfinavir mesylate
Drug: Efavirenz

SUMMARY:
Indinavir is usually taken three times a day. The purpose of this study is to see if it is safe and effective to take indinavir only twice a day plus nelfinavir (also taken twice a day) and efavirenz (taken once a day).

DETAILED DESCRIPTION:
Patients receive a treatment regimen consisting of nelfinavir, indinavir, and efavirenz for 48 weeks. During the study, patients are evaluated for changes from baseline in plasma HIV-1 RNA levels and lymphocyte subsets and for development of adverse events and toxicities. After Week 48, patients with documented virologic response are eligible to continue receiving study treatments and to attend scheduled follow-up visits. Patients who experience virologic failure are discontinued from the study.

ELIGIBILITY:
Inclusion Criteria

You may be eligible for this study if you:

* Are HIV-positive.
* Are at least 13 years old (consent of parent or guardian required if under 18).
* Have a viral load of at least 10,000 copies/ml within 30 days of study entry.
* Agree to use a barrier method of birth control, such as condoms, during the study.

Exclusion Criteria

You will not be eligible for this study if you:

* Have hepatitis.
* Have any other serious medical condition besides HIV infection.
* Are allergic to indinavir, nelfinavir, or efavirenz.
* Have ever taken NNRTIs or protease inhibitors.
* Have had chemotherapy or radiation therapy within 30 days of study entry. (Local radiation therapy is allowed.)
* Have taken certain other medications that might affect your immune system such as interleukin-2, interferon, or a vaccine within 30 days of study entry.
* Are enrolled or plan to enroll in another anti-HIV drug study during this study.
* Are pregnant or breast-feeding.
* Abuse alcohol or drugs.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 6

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Pacific Oaks Med Group, Beverly Hills, California
  - Univ of Colorado / Health Science Ctr, Denver, Colorado
  - AIDS Research Consortium of Atlanta, Atlanta, Georgia
  - Brown Univ School of Medicine, Providence, Rhode Island
  - Hampton Roads Med Specialists, Hampton, Virginia